CLINICAL TRIAL: NCT01292993
Title: A Phase 1, Randomized, Open-Label, 3-Period, 3-Treatment, Single-dose Crossover Study to Evaluate the Pharmacokinetic Interaction of LX4211 and Metformin in Healthy Subjects
Brief Title: A Study to Evaluate the Interaction of LX4211 and Metformin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Ikenna Ogbaa, MD, Lexicon Pharmaceuticals, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LX4211.1-103-DDI; LX4211.103 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2011-02-08; First posted 2011-02-10 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): 400 mg LX4211
  Interventions: Drug: 400 mg LX4211
- Treatment B (Experimental): 1000 mg metformin
  Interventions: Drug: 1000 mg metformin
- Treatment C (Experimental): 400 mg LX4211 + 1000 mg metformin
  Interventions: Drug: 400 mg LX4211; Drug: 1000 mg metformin

INTERVENTIONS:
Drug: 400 mg LX4211 — 400 mg of LX4211 given as a solid oral dose form
  Arms: Treatment A; Treatment C
Drug: 1000 mg metformin — 1000 mg metformin given as a solid oral dose form
  Arms: Treatment B; Treatment C

SUMMARY:
The purpose of this study is to determine the effects of LX4211 and metformin on each other when given at the same time as single doses to healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 to ≤55 years of age. Females must be of non-childbearing potential.
* Body mass index (BMI)≥18 to ≤35 kg/sq m
* Able to provide written consent
* Vital signs within sponsor-defined ranges

Exclusion Criteria:

* Use of any medication, including any prescription, over-the-counter, herbal tea, or other supplements within 5 days of dosing
* No investigational agent or study treatment within 30 days prior to Day 1.
* No protein or antibody-based therapeutic agents within 3 months prior to screening
* Use of any tobacco product
* History of bariatric surgery or any gastrointestinal surgery that may induce malabsorption
* History of any major surgery within 6 months prior to screening
* History of any serious adverse reaction or hypersensitivity to metformin or LX4211.
* History of renal disease or significantly abnormal kidney function test
* History of hepatic disease or significantly abnormal liver function test
* History of any active infection within 30 days prior to Day 1
* History of any surgical or medical condition or clinically significant laboratory or physical finding
* Positive urine glucose at Screening
* Use of drugs or alcohol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of LX4211 and metformin after concurrent single-dose administration | Up to 43 days, including screening

SECONDARY OUTCOMES:
Urinary glucose excretion | Up to 43 days, including screening
Fasting plasma glucose | Up to 43 days, including screening
Postprandial glucose | Up to 43 days, including screening
Insulin | Up to 43 days, including screening
Peptide YY | Up to 43 days, including screening
Glucagon-like peptide (GLP-1) | Up to 43 days, including screening
Glucose-dependent insulinotropic peptide | Up to 43 days, including screening

CONTACTS AND LOCATIONS:
Overall Officials: Ikenna Ogbaa, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, San Antonio, Texas, United States